CLINICAL TRIAL: NCT04721483
Title: Selective T3-T4 Sympathicotomy Versus Gray Ramicotomy on Outcome and Quality of Life in Hyperhidrosis Patients. A Randomized Clinical Trial
Brief Title: T3-T4 Gray Sympathycotomy Versus Ramicotomy for Hyperhidrosis
Acronym: T3-T4RY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEIm 24-02-2016
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Hyperhidrosis; Compensatory Sweating; Compensatory Hyperhidrosis
Keywords: Hyperhidrosis; Ramicotomy; Sympathectomy; Sympathicotomy; Compensatory hyperhidrosis; Gustatory sweating
MeSH Terms: conditions — Hyperhidrosis; Sweating, Gustatory

STUDY DESIGN:
Intervention Model Description: Two groups. One with T3-T4 sympathicotomy and another with T3-T4 gray ramicotomy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients distributed in a prospective randomized fashion between two groups. We calculated the sample size based on previous research and used a block randomization model. We took eight blocks of four and two blocks of five patients with a random distribution of two patients from each group. This project was blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T3-T4 sympathicotomy (Active Comparator): In this group, patients underwent a classical T3 and T4 sympathicotomy to treat primary palmar hyperhidrosis
  Interventions: Procedure: Ramicotomy
- T3-T4 ramicotomy (Experimental): In this group, patients underwent a selective T3 and T4 gray ramicotomy
  Interventions: Procedure: Ramicotomy

INTERVENTIONS:
Procedure: Ramicotomy — We will selectively lesion the gray rami communicantes from T3 and T4 thoracic sympathetic ganglia

SUMMARY:
It is presented a further refinement in palmar hyperhidrosis's surgical treatment to improve results and reduce side effects, mainly compensatory hyperhidrosis. It seems that a more selective sympathetic system lesion, namely a selective T3 and T4 gray rami communicantes lesion, allows retaining some residual sweating in the hands without inducing compensatory sweating in the abdomen, thighs, and feet. The result is greater patient satisfaction. There has been a long journey since Wittmosser et al. suggested the technique of gray and white ramicotomy in 1992. In this way, the attending physicians have refined the surgical procedure progressively. The two last research groups reporting their results with selective gray ramicotomy (the idea now is not to lesion the white rami communicantes) entailed extensive lesions (T2 to T4/T5). This study shows that a more selective T3 and T4 selective gray ramicotomy achieves excellent results with fewer side effects. Thus, it is a further step toward improving outcomes, reducing side effects, and increasing patients' satisfaction.

Additionally, the present work has concentrated on objective ways to measure compensatory hyperhidrosis by measuring the sweat production in milliliters of water and the temperature changes in degrees Celsius. This accurate measurement removes the subjectivity induced when we base the results on the treating physicians' opinions or the patients themselves.

The objective measurement of the sweat production in milliliters of water and temperature rise in degrees Celsius has allowed the research group to reach conclusions independent of opinions both from treating physicians and patients themselves. Also, a more selective gray rami communicantes lesion can achieve better results with less compensatory hyperhidrosis and with better patient's satisfaction

DETAILED DESCRIPTION:
Ever since the introduction of thoracic sympathectomy in the treatment of palmar and axillary hyperhidrosis, there has been a continuous quest to find a way to reduce its most unpleasant side effect: compensatory hyperhidrosis (CH). Following the idea of minimizing the surgically induced damage to the sympathetic chain, Wittmoser introduced in 1992, the ramicotomy technique. It entailed the selective lesion of the rami communicantes, both white and gray, from T2 to T4-T5. This surgical technique was not as selective as expected because it damaged the sympathetic input for the lungs and heart, and the head and face. Wittmoser described this surgical technique but never published any results. Gossot4 in 1997 compared this technique with the sympathectomy of the same ganglia in 54 patients. He found that CH's incidence was the same in both groups, but the severity was less in the ramicotomy than in the sympathectomy group. The recurrence rate was more prominent in the first than in the second group (5% ramicotomy versus 0% sympathectomy). Other researchers have confirmed these results.

More studies compared the sympathectomy with the ramicotomy in the following years, confirming that ramicotomy has a lower incidence of CH5-10, with less dry hands but with some recurrences.

In a step forward, Coveliers et al.11 lesioned only the T2 T3 and T4 gray rami communicantes, not touching the sympathetic chain or the white rami communicantes, with CH dropping to 7.2% and no recurrences. Akil et al.12 reported the lesion of the T2-T5 gray rami communicantes with no CH and again with no recurrences. Both studies entail a more extensive lesion, including T2, and one of those studies, T5. There is an agreement to avoid lesioning T2 in many previous reports to reduce the incidence and severity of CH.

ELIGIBILITY:
Inclusion Criteria:

* palmar HH with or without axillary HH refractive to conservative treatments
* or reluctant to continue with them after six months and willing to undergo surgical treatment,
* Hyperhidrosis Disease Severity Score grade D

Exclusion Criteria:

* previous thoracic pathology (lung infections, particularly pulmonary empyema, pneumothorax, hemothorax, rib fractures, neoplasms)
* heart failure
* hypothyroidism
* tuberculosis
* bradycardia (40 pulsations/min)
* alcoholism
* drug addiction
* BMI >30
* pregnancy
* generalized HH or related to any health disorder
* comorbidities
* or medication intake that induces excessive sweating
* patients with primary facial or plantar HH
* patients not complying with follow-ups

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Compensatory sweating | 1 year
  We will measure the increase in sweating in the chest, abdomen thighs and feet by capturing the sweat produced in these body areas in a period of 15 minutes in a closed room at 25ºC and 85% humidity. The sweat will be captured with a special cellulose pad and these pads will be weighted with a precision scale before and after being placed in the body areas to be analysed. The sweat production will be known by the milliliters of water captured in the pads used to capture it
Postoperative quality of life | 1 year
  We will compare with a questionnaire that patients will fulfill baseline and in every follow-up visit on the quality of life. It will be used the quality of life questionnaire developed by Amir M, Arish A, Weinstein Y, Pfeffer M, Levy Y. Impairment in quality of life among patients seeking surgery for hyperhidrosis (excessive sweating): preliminary results. Isr J Psychiatry Relat Sci. 2000;37(1):25-31.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital General Universitario de Valencia, Valencia
  - Vicente Vanaclocha, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gossot D, Toledo L, Fritsch S, Celerier M. Thoracoscopic sympathectomy for upper limb hyperhidrosis: looking for the right operation. Ann Thorac Surg. 1997 Oct;64(4):975-8. doi: 10.1016/s0003-4975(97)00799-6. PMID 9354512
- [Background] Cho HM, Chung KY, Kim DJ, Lee KJ, Kim KD. The comparison of VATS ramicotomy and VATS sympathicotomy for treating essential hyperhidrosis. Yonsei Med J. 2003 Dec 30;44(6):1008-13. doi: 10.3349/ymj.2003.44.6.1008. PMID 14703609
- [Background] Lee DY, Kim DH, Paik HC. Selective division of T3 rami communicantes (T3 ramicotomy) in the treatment of palmar hyperhidrosis. Ann Thorac Surg. 2004 Sep;78(3):1052-5. doi: 10.1016/j.athoracsur.2004.03.034. PMID 15337046
- [Background] Cheng YJ, Wu HH, Kao EL. Video-assisted thoracoscopic sympathetic ramicotomy for hyperhidrosis--a way to reduce the complications. Ann Chir Gynaecol. 2001;90(3):172-4. PMID 11695787
- [Background] Lee DY, Paik HC, Kim DH, Kim HW. Comparative analysis of T3 selective division of rami communicantes (ramicotomy) to T3 sympathetic clipping in treatment of palmar hyperhidrosis. Clin Auton Res. 2003 Dec;13 Suppl 1:I45-7. doi: 10.1007/s10286-003-1115-1. PMID 14673673
- [Background] Kim DY, Paik HC, Lee DY. Comparative analysis of T2 selective division of rami-communicantes (ramicotomy) with T2 sympathetic clipping in the treatment of craniofacial hyperhidrosis. Eur J Cardiothorac Surg. 2004 Aug;26(2):396-400. doi: 10.1016/j.ejcts.2004.04.030. PMID 15296904
- [Background] Hwang JJ, Kim DH, Hong YJ, Lee DY. A comparison between two types of limited sympathetic surgery for palmar hyperhidrosis. Surg Today. 2013 Apr;43(4):397-402. doi: 10.1007/s00595-012-0246-1. Epub 2012 Jul 15. PMID 22798011
- [Background] Coveliers H, Meyer M, Gharagozloo F, Wisselink W, Rauwerda J, Margolis M, Tempesta B, Strother E. Robotic selective postganglionic thoracic sympathectomy for the treatment of hyperhidrosis. Ann Thorac Surg. 2013 Jan;95(1):269-74. doi: 10.1016/j.athoracsur.2012.08.013. Epub 2012 Nov 14. PMID 23158099
- [Background] Akil A, Semik M, Fischer S. Efficacy of Miniuniportal Video-Assisted Thoracoscopic Selective Sympathectomy (Ramicotomy) for the Treatment of Severe Palmar and Axillar Hyperhidrosis. Thorac Cardiovasc Surg. 2019 Aug;67(5):415-419. doi: 10.1055/s-0038-1642030. Epub 2018 May 8. PMID 29739022
- [Background] Zhang W, Yu D, Wei Y, Xu J, Zhang X. A systematic review and meta-analysis of T2, T3 or T4, to evaluate the best denervation level for palmar hyperhidrosis. Sci Rep. 2017 Mar 9;7(1):129. doi: 10.1038/s41598-017-00169-w. PMID 28273934
- [Background] Cai SW, Shen N, Li DX, Wei B, An J, Zhang JH. Compensatory sweating after restricting or lowering the level of sympathectomy: a systematic review and meta-analysis. Clinics (Sao Paulo). 2015 Mar;70(3):214-9. doi: 10.6061/clinics/2015(03)11. Epub 2015 Mar 1. PMID 26017654
- [Background] Scognamillo F, Serventi F, Attene F, Torre C, Paliogiannis P, Pala C, Trignano E, Trignano M. T2-T4 sympathectomy versus T3-T4 sympathicotomy for palmar and axillary hyperhidrosis. Clin Auton Res. 2011 Apr;21(2):97-102. doi: 10.1007/s10286-010-0110-6. Epub 2011 Jan 19. PMID 21243401
- [Background] Dogru MV, Sezen CB, Girgin O, Cansever L, Kocaturk CI, Metin M, Dincer SI. Is there any relationship between quality of life and the level of sympathectomy in primary palmar hyperhidrosis? Single-center experience. Gen Thorac Cardiovasc Surg. 2020 Mar;68(3):273-279. doi: 10.1007/s11748-019-01210-7. Epub 2019 Sep 21. PMID 31542862
- [Background] Weksler B, Blaine G, Souza ZB, Gavina R. Transection of more than one sympathetic chain ganglion for hyperhidrosis increases the severity of compensatory hyperhidrosis and decreases patient satisfaction. J Surg Res. 2009 Sep;156(1):110-5. doi: 10.1016/j.jss.2009.04.015. Epub 2009 May 14. PMID 19631343
- [Background] Yazbek G, Wolosker N, de Campos JR, Kauffman P, Ishy A, Puech-Leao P. Palmar hyperhidrosis--which is the best level of denervation using video-assisted thoracoscopic sympathectomy: T2 or T3 ganglion? J Vasc Surg. 2005 Aug;42(2):281-5. doi: 10.1016/j.jvs.2005.03.041. PMID 16102627
- [Result] WITTMOSER R. [Thoracoscopic sympathicotomy in circulation disorders of the arm]. Langenbecks Arch Klin Chir Ver Dtsch Z Chir. 1959;292:318-23. No abstract available. German. PMID 13845515